CLINICAL TRIAL: NCT00172419
Title: Statin-Induced Vulnerable Plaque Regression After Atorvastatin Treatment: Serial Evaluation by 18F-Fluorodeoxyglucose Positron Emission Tomography Study
Brief Title: The Effects of Atorvastatin on Vulnerable Plaques in Untreated Dyslipidemic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Pfizer (Industry)
Responsible Party: Wei-Shiung Yang, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 931204
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: Hyperlipidemia
Keywords: statin, inflammation, FDG, positron emission tomography
MeSH Terms: conditions — Hyperlipidemias; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin, 40 mg/day for 12 weeks
  Other Names: Atorvastatin (Lipitor, 40mg)

SUMMARY:
Inflammation is important in the both pathogenesis and outcome of atherosclerosis. Plaques containing numerous inflammatory cells, particular macrophages, have a high risk of rupture.We hypothesize that statin-induced plaque regression could be monitored clinically by use of FDG PET/CT approach, and can be detected noninvasively earlier than previously reported.

DETAILED DESCRIPTION:
Cardiovascular events are the leading cause of death in developed countries worldwide, including Taiwan. The disruption of atherosclerotic plaques and the subsequent formation of thrombi are currently recognized as the major cause of morbidity and mortality of cardiovascular diseases. Therefore, early detection of vulnerable plaques is clinically important for risk stratification and also to provide early treatment. Several imaging approaches have been adapted to detect vulnerable plaques, including conventional X-ray contrast angiography, catheter capable of detecting temperature heterogeneity, infrared light or pH heterogeneity, ultrasonography (including intravascular ultrasound), high-resolution computed tomography and MRI. However, most of them are based on morphologic characteristics of atheroma. Moreover, although statin-induced lipid lowering and clinical benefits may occur in a matter of weeks, stain-mediated plaque volume regression has been measured in terms of years after the initiation of statin therapy. These discrepancies highlight the need for greater insight into the mechanisms and time course of statin-induced plaque regression.

As we know, inflammation may play a significant role in the pathogenesis and progression of atherosclerosis and subsequent vulnerable plaque rupture. Recently, 18F-fluorodeoxyglucose (FDG) positron emission tomography (PET), by use of 18FDG taken up by surrounding macrophages and smooth muscle cells, has been reported to detect atherosclerotic lesions by bio-pathologic functions. More and more evidence showed that FDG uptake is a marker of hypermetabolic state of atheromatous plaques, which is related to dense cellular infiltrate, and contributes to the identification of a subgroup of patients at high risk of complications. Recently, a combined PET/CT is emerged as a promising modality and is now beginning to be used more routinely in clinical situation, providing better localization and detecting calcification at the same time. Therefore, the use of FDG PET/CT might be a more sensitive and quantification method to monitor the inflammatory activity of vulnerable plaque after aggressive statin treatment. It could also provide the mechanism of early beneficial effects of statin treatment.

Our subject is to investigate prospectively the statin effects of lipid lowering and anti-inflammatory on human atherosclerotic lesions. We hypothesize that statin-induced plaque regression could be monitored clinically by use of FDG PET/CT approach, and can be detected noninvasively earlier than previously reported, and providing information of early statin efficacy caused by stabilization of vulnerable plaque without affecting the lumen size.

ELIGIBILITY:
Inclusion Criteria: Untreated dyslipidemic (LDL cholesterol >110 mg/dl) subjects with documented atherosclerosis in at least 1 vascular territory: at least moderate (≧4.0mm) aortic atherosclerosis by transesophageal echocardiography or CT/MRI, angiographically documented with coronary artery stenosis (≧50% luminal stenosis), ultrasonographically documented significant extracranial arterial stenosis (≧50%), history of ischemic stroke and transient ischemic attack (TIA), or documented peripheral vascular disease. Exclusion Criteria: Acute illness,infection, inflammation or major systemic diseases, T-Bil >3 mg/dl, or Creatinine >3 mg/dl.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Plaque location and activity at baseline, and compare with the follow-up scans site by site. | 12 w

SECONDARY OUTCOMES:
Lipid profile | 12 w
Biomarkers | 12 w

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Shiung Yang, MD, phD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang YY, Wu YW, Lee JK, Lin YM, Lin YT, Kao HL, Hung CS, Lin HJ, Lin YH. Effects of 12 weeks of atorvastatin therapy on myocardial fibrosis and circulating fibrosis biomarkers in statin-naive patients with hypertension with atherosclerosis. J Investig Med. 2016 Oct;64(7):1194-9. doi: 10.1136/jim-2016-000092. Epub 2016 Jul 18. PMID 27430242